CLINICAL TRIAL: NCT03829046
Title: The Effects of Evolocumab on Endothelial and Inflammatory Biocellular Markers in Patients With Diabetes and Atherosclerotic Vascular Disease (METCHNIKOFF)
Brief Title: The Effects of Evolocumab in Patients With Diabetes and Atherosclerotic Vascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Robert Rosenson (Other)
Collaborators: Amgen (Industry); University of Toronto (Other); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Robert Rosenson, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GCO 18-1412; 20167719 (Other: Amgen)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Atherosclerotic Vascular Disease; Type2 Diabetes; Microvascular Dysfunction
Keywords: PCSK9 inhibition; Evolocumab; Inflammatory Signals; Circulating monocyte subsets
MeSH Terms: conditions — Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: A multi-center, double-blind, randomized, placebo-controlled, parallel group Phase IV study with two treatment arms: evolocumab SC 420 mg/dL QM or matching placebo. The identity of the treatments will be concealed by the use of matching placebo to the study drug that are identical in packaging, labeling, appearance and schedule of administration.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The identity of the treatments will be concealed by the use of matching placebo to the study drug that are identical in packaging, labeling, appearance and schedule of administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo SC QM
  Interventions: Drug: Placebo
- Evolocumab (Active Comparator): Evolocumab SC 420mg/dL QM
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Placebo — 12 weeks of treatment
  Arms: Placebo
Drug: Evolocumab — 12 weeks of treatment
  Arms: Evolocumab

SUMMARY:
Experimental models have linked lipid lowering therapies with systemic inflammation; however, relatively little is known about this network in clinical populations and specifically how it changes with PCSK9 inhibition. The eligible subjects will have 6 visits in 13 to 16 weeks and will have Repatha/placebo 140mg subcutaneous every 4 weeks for 3 times since randomization visit, blood tests will be done in each visit to evaluate the effects of evolocumab upon biocellular markers potentially altered by PCSK9 inhibition in a population of type 2 diabetes patients with microvascular dysfunction.

Primary Aims:

Determine the ACUTE and SHORT-TERM effects of PCSK9 inhibition with evolocumab on biocellular markers of inflammation, immune mediated thrombosis and rheology. The data from this trial will be used to support a clinical trial to assess the role of PCSK9 inhibition in type 2 diabetes patients with cardiac microvascular dysfunction.

Secondary Aims:

1. To define the association between PCSK 9 concentrations and immune-related phenotype.
2. To define the association between Lp(a) concentrations, oxidized phospholipids (OxPL), ApoB, biocellular markers of inflammation, tissue factor and immunothrombosis.

DETAILED DESCRIPTION:
Multi-center, double-blind, randomized, placebo-controlled, parallel group Phase IV study with two treatment arms: evolocumab SC 420 mg/dL QM or matching placebo. The population will include 40 participants with documented Atherosclerotic Vascular Disease (CAD, Stroke, PAD) and type 2 diabetes who receive treatment with maximal tolerated statin therapy and stable doses of anti-hyperglycemic therapy.

Subjects will be followed for 12 weeks during the treatment phase, maintaining the double-blind throughout. Assessments of ACUTE and SHORT-TERM effects of PCSK9 inhibition with evolocumab on biocellular markers of endothelial function will be measured at baseline, Week 2, and Week 12. Safety assessments will be undertaken at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age signing of informed consent;
* A history of clinical ASCVD, which is defined as: acute coronary syndrome, or a history of MI, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack (TIA), or peripheral arterial disease presumed to be of atherosclerotic origin;
* Clinical diagnosis of type 2 diabetes according to ADA/ CDA guidelines;
* Subject on stable dose of maximally-tolerated statin therapy for ≥4 weeks prior to screening and LDL-c ≥70mg/dL. For subjects whose maximally tolerated dose of statin is no type or dose (i.e. determined to be statin intolerant by primary investigator), background lipid-lowering therapy is not required;
* Fasting triglycerides ≤400mg/dL (4.52mmol/L) by central laboratory at screening;
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures;
* Abnormal urinary Albumin Creatinine Ratio (ACR) as defined by an ACR ≥2;
* Subject tolerates screening placebo injection.

Exclusion Criteria:

* Personal or family history of hereditary muscular disorders;
* NYHA III or IV heart failure, or last know left ventricular ejection fraction (LVEF) <30%;
* Uncontrolled serious cardiac arrhythmia defined as recurrent and highly symptomatic ventricular tachycardia, atrial fibrillation with rapid ventricular response, or supraventricular tachycardia that are not controlled by medications, in the past 6 weeks prior to randomization;
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery graft (CABG) or stroke within 3 months prior to randomization;
* Planned cardiac surgery or revascularization;
* Moderate to severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <30mL/min/1.73m2 at screening;
* Type 1 diabetes, poorly controlled type 2 diabetes (HbA1c >10%), newly diagnosed type 2 diabetes (within 6 months of randomization), or laboratory evidence of diabetes during screening (fasting serum glucose ≥126mg/dL [7.0mmol/L] or HbA1c ≥6.5% without prior diagnosis of diabetes;
* Uncontrolled hypertension, defined as sitting systolic blood pressure (SBP) >160mmHg or diastolic BP (DBP) >100mmHg;
* Subject who has taken a cholesterol easter transfer protein (CETP) inhibitor in the last 12 months prior to LDL-c screening, such as: anacetrapib, dalcetrapib or evacetrapib;
* Treatment in the last 3 months prior to LDL-c screening with any of the following drugs: systemic cyclosporine, systemic steroids (e.g. IV, intramuscular [IM], or PO) (Note: hormone replacement therapy is permitted), vitamin A derivatives and retinol derivatives for the treatment of dermatologic conditions (e.g. Accutane); (Note: vitamin A in a multivitamin preparation is permitted). Topical retinol prescription and non-prescription derivatives or creams are permitted;
* Uncontrolled hypothyroidism or hyperthyroidism as defined by thyroid stimulating hormone (TSH) <1.0 time the lower limit of normal or >1.5 times the ULN, respectively, at screening. Potential subjects with TSH <1.0 time the lower limit of normal due to thyroid replacement therapy is not considered an exclusion;
* Active liver disease or hepatic dysfunction, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the ULN as determined by central laboratory analysis at screening;
* Known active infection or major hematologic, renal metabolic, gastrointestinal or endocrine dysfunction in the judgment of the investigator;
* Diagnosis of deep vein thrombosis or pulmonary embolism within 3 months prior to randomization;
* Unreliability as a study participant based on the investigator's (or designee's) knowledge of the subject (e.g. alcohol or other drug abuse);
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s);
* Female subject who has either (1) not used at least 1 highly effective method of contraception for at least 1 month prior to screening or (2) is not willing to use such a method during treatment and for an additional 15 weeks after the end of treatment, unless the subject is sterilized or postmenopausal;
* Subject who is pregnant or breast feeding, or planning to become pregnant during treatment and/ or within 15 weeks after the end of treatment;
* Use of PCSK9 inhibitor within 10 weeks from screening;
* Subject who has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures;
* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years;
* Subject who has known sensitivity to any of the products or components to be administered during dosing;
* Subject who is likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge;
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the principal investigator would pose a risk to subject or interfere with the study evaluation, procedures or completion;
* Blood donation 4 weeks prior to screening, or stated intention to donate blood or blood products during the period of the study or within one month following completion of the study;
* Subjects who have participated in other studies within 30 days prior to screening, or have five times the plasma half-life (if known) of the investigational drug, whichever is longer;
* BMI>40kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both: male and female
Enrollment: 41 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rosenson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kim A Connelly, MD, Principal Investigator — St. Michael's Hospital at University of Toronto
Locations (2):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- St. Michael's - University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilot study and all data from this trial will be used to support a bigger clinical trial to assess the role of PCSK9 inhibition in type 2 diabetes patients with cardiac microvascular dysfunction.

REFERENCES:
- [Background] Tall AR, Yvan-Charvet L. Cholesterol, inflammation and innate immunity. Nat Rev Immunol. 2015 Feb;15(2):104-16. doi: 10.1038/nri3793. PMID 25614320
- [Background] Chatzizisis YS, Coskun AU, Jonas M, Edelman ER, Feldman CL, Stone PH. Role of endothelial shear stress in the natural history of coronary atherosclerosis and vascular remodeling: molecular, cellular, and vascular behavior. J Am Coll Cardiol. 2007 Jun 26;49(25):2379-93. doi: 10.1016/j.jacc.2007.02.059. Epub 2007 Jun 8. PMID 17599600
- [Background] Dai G, Kaazempur-Mofrad MR, Natarajan S, Zhang Y, Vaughn S, Blackman BR, Kamm RD, Garcia-Cardena G, Gimbrone MA Jr. Distinct endothelial phenotypes evoked by arterial waveforms derived from atherosclerosis-susceptible and -resistant regions of human vasculature. Proc Natl Acad Sci U S A. 2004 Oct 12;101(41):14871-6. doi: 10.1073/pnas.0406073101. Epub 2004 Oct 4. PMID 15466704
- [Background] Traub O, Berk BC. Laminar shear stress: mechanisms by which endothelial cells transduce an atheroprotective force. Arterioscler Thromb Vasc Biol. 1998 May;18(5):677-85. doi: 10.1161/01.atv.18.5.677. PMID 9598824
- [Background] Nahrendorf M, Pittet MJ, Swirski FK. Monocytes: protagonists of infarct inflammation and repair after myocardial infarction. Circulation. 2010 Jun 8;121(22):2437-45. doi: 10.1161/CIRCULATIONAHA.109.916346. No abstract available. PMID 20530020
- [Background] Chang HN, Leroueil PR, Selwa K, Gasper CJ, Tsuchida RE, Wang JJ, McHugh WM, Cornell TT, Baker JR Jr, Goonewardena SN. Profiling inflammatory responses with microfluidic immunoblotting. PLoS One. 2013 Nov 27;8(11):e81889. doi: 10.1371/journal.pone.0081889. eCollection 2013. PMID 24312374
- [Derived] Rosenson RS, Tate A, Mar P, Grushko O, Chen Q, Goonewardena SN. Inhibition of PCSK9 with evolocumab modulates lipoproteins and monocyte activation in high-risk ASCVD subjects. Atherosclerosis. 2024 May;392:117529. doi: 10.1016/j.atherosclerosis.2024.117529. Epub 2024 Mar 25. PMID 38583289
- See also: Inflammation in atherosclerosis — https://www.nature.com/articles/nature01323
- See also: Hemodynamic Shear Stress via ROS Modulates PCSK9 Expression in Human Vascular Endothelial and Smooth Muscle Cells and Along the Mouse Aorta. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4361218/
- See also: Local effects of human PCSK9 on the atherosclerotic lesion. — https://www.ncbi.nlm.nih.gov/pubmed/26333678

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo SC QM x 12 weeks of treatment
- Evolocumab: Evolocumab SC 420mg/dL QM x 12 weeks of treatment
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 20 | 21
Completed | 19 | 21
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.3) | 65.9 (7.7) | 65.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 17
  Not Hispanic or Latino | 8 | 15 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 9 | 20
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking [Count of Participants; unit: Participants]
  Current | 5 | 2 | 7
  Former | 9 | 9 | 18
  Never smoker | 5 | 10 | 15
Diabetes [Count of Participants; unit: Participants] | 19 | 21 | 40
Hypertension [Count of Participants; unit: Participants] | 17 | 21 | 38
Cardiovascular Disease (CVD) [Count of Participants; unit: Participants]
  Coronary Artery Disease (CAD) | 11 | 15 | 26
  Carotid Disease | 2 | 2 | 4
  Peripheral Artery Disease (PAD) | 6 | 4 | 10
Family History [Count of Participants; unit: Participants]
  Premature CAD | 4 | 2 | 6
  No premature CAD | 15 | 19 | 34
Medication Use [Count of Participants; unit: Participants]
  Antihypertensive | 17 | 21 | 38
  Antidiabetics | 18 | 20 | 38
  High intensity Statins | 11 | 12 | 23
  Low to moderate intensity Statins | 6 | 5 | 11
  No Statin (Statin intolerance) | 2 | 4 | 6
Cholesterol Panel [Mean (Standard Deviation); unit: mg/dL] — Total Cholesterol, Low-density Lipoprotein - cholesterol (LDL-C), High-density Lipoprotein - cholesterol (HDL), Triglycerides (TG)
  mg/dL
    Total Cholesterol | 189.9 (39.1) | 180.0 (34.7) | 184.7 (36.2)
    LDL-C | 114.2 (30.4) | 107.7 (32.0) | 110.8 (30.6)
    HDL | 51.6 (17.8) | 44.9 (11.9) | 48.1 (15.0)
    Triglycerides | 129.2 (56.0) | 145.0 (59.2) | 137.5 (56.8)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.4 (0.3) | 4.4 (0.3) | 4.4 (0.3)
Fibrinogen [Mean (Standard Deviation); unit: mg/dL] | 329.9 (80.6) | 317.5 (131.1) | 323.4 (107.5)
HbA1c (glycated hemoglobin) [Mean (Standard Deviation); unit: percentage of hgb coated with glucose] | 7.0 (1.2) | 7.0 (1.1) | 7.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety as measured by number of adverse events, defined as any untoward medical occurrence in a subject who has been administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: up to 12 weeks
Measure: Number; unit: events
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 19 | 21
events | 13 | 13

2. Secondary Outcome: Seattle Angina Questionnaire
Description: The Seattle Angina Questionnaire is a quality-of-life measure for patients with coronary artery disease. The SAQ is a self-report instrument with 19 items that yields five subscale scores: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life. There is no summary score generated.
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: MDA Level
Description: Malondialdehyde levels to measure oxidative stress
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: MPO Level
Description: Myeloperoxidase level to measure inflammation
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: IL-6 Level
Description: Interleukin-6 levels to measure cytokines
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: IL-18 Level
Description: Interleukin-8 levels to measure cytokines
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: TNF-α Level
Description: Tumor necrosis factor alpha levels to measure cytokines
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: PECAM Level
Description: Platelet endothelial cell adhesion molecule levels to measure vascular endothelial activation
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: ICAM Level
Description: Intercellular adhesion molecule levels to measure vascular endothelial activation
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: VCAM Level
Description: Vascular cell adhesion molecule levels to measure vascular endothelial activation
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Alpha5/Beta3 Activation Levels
Description: Alpha 5/Beta 3 levels to measure vascular endothelial activation
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/19 | 4/21
Other Adverse Events (participants affected / at risk) | 10/19 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Evolocumab (N=21)
Acute Osteomyelitis (Infections and infestations) | 0 | 1
Seizure Type activity (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Critical limb ischemia (Vascular disorders) | 1 | 0
Exertional Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hospital Admission- Unsuccessful PTA (Cardiac disorders) | 1 | 0
Cervical Stenosis of Spine (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Evolocumab (N=21)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Flu-like Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin itching (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest Pain (Cardiac disorders) | 2 | 2
pinch at injection site when consumes greasy food (Skin and subcutaneous tissue disorders) | 1 | 0
weird taste in mouth right after injection (General disorders) | 0 | 1
pain under breast on and off (Skin and subcutaneous tissue disorders) | 0 | 1
patient felt disoriented and confused after first injection (General disorders) | 1 | 0
worsening memory (Psychiatric disorders) | 1 | 0
drowsy right after injections (General disorders) | 1 | 0
stomach cramps (General disorders) | 1 | 0
reduced appetite (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03829046/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03829046/ICF_001.pdf